CLINICAL TRIAL: NCT05608642
Title: Comparison of the Efficiency of Intravenous Treatments Used in Bridge Treatment of Medication Overuse Headache
Brief Title: Intravenous Treatments Used in Medication Overuse Headache Bridge Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Director, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Medication Overuse Headache
Record Dates: First submitted 2022-10-23; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Medication Overuse Headache
Keywords: lidocaine; prednisolone; intravenous hydration
MeSH Terms: conditions — Headache Disorders, Secondary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group given intravenous hydration (Active Comparator): The first group consists of patients given 500 cc intravenous saline for 1 hour.
  Interventions: Other: Intravenous hydration
- Group given intravenous prednisolone (Active Comparator): Second group; consists of patients who were given 80 mg of intravenous prednisolone for the first 4 days and then given gradually decreasing doses of prednisolone in the following days.
  Interventions: Other: Intravenous prednisolone
- Group given intravenous lidocaine (Active Comparator): Third group; includes patients given 2 mg/kg intravenous lidocaine by 1-hour infusion.
  Interventions: Other: Intravenous lidocaine

INTERVENTIONS:
Other: Intravenous hydration — 500 cc intravenous serum for 1 hour in the first group service consists of patients who have been given.
  Arms: Group given intravenous hydration
Other: Intravenous prednisolone — The second group consisted of patients who were given 80 mg intravenous prednisolone for the first 4 days and then gradually reduced doses of prednisolone in the following days.
  Arms: Group given intravenous prednisolone
Other: Intravenous lidocaine — The third group includes patients in whom 2 mg/kg of intravenous lidocaine is given by 1-hour infusion.
  Arms: Group given intravenous lidocaine

SUMMARY:
Medication overuse headache is the chronicity of headaches, which occurs more than 15 days a month, as a result of frequent use of painkillers, opioids or migraine attack drugs (ergotamine, triptan) in individuals with pre-existing primary headache disease.

In the treatment of this headache, two ways can be followed as slow drug discontinuation or sudden drug discontinuation. The most commonly used method is the sudden discontinuation of the overused analgesic agent, the initiation of prophylactic treatment, and then the application of bridge therapy for 6-10 days. Intravenous hydration, steroids, antiemetics, neuroleptic drugs and local anesthetic drugs such as lidocaine can be used in bridge treatment.

DETAILED DESCRIPTION:
In our clinic, we routinely apply intravenous 1.5 mg/kg lidocaine, intravenous prednisolone and intravenous saline treatments as bridge treatment to patients diagnosed with medication overuse headache. In this study, we aimed to compare the efficacy of intravenous lidocaine, intravenous steroids and intravenous hydration therapy, which were used as bridge therapy after the cessation of analgesic use in patients with medication overuse headache.

Patients who applied to the algology outpatient clinic and who were diagnosed with drug overuse headache and treated were evaluated by dividing them into 3 different groups. It was planned to include 15 patients in each group. The first group consists of patients who were given 500 cc of intravenous saline for 1 hour in the service. The second group consisted of patients who were given 80 mg intravenous prednisolone for the first 4 days and then gradually reduced doses of prednisolone in the following days. The third group includes patients in whom 2 mg/kg intravenous lidocaine was administered as a 1-hour infusion, monitored in the ward.

Pain intensity will be evaluated by visual analog scale (VAS) in all patients after treatment, at 1 month and 3 months. In addition, the number of days with pain and the number of analgesics used in the 3-month period after the end of the treatment will be evaluated and the Quality of Life Scale will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Medication overuse headache
* Chronic migraine

Exclusion Criteria:

* Other headaches will not accompany (tension-type headache, cluster...)
* Pregnancy
* Epilepsia
* Heart disease
* Bradikardia
* Hypertension
* Diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 4 weeks
  It is a scale that measures the severity of pain. Scored between ''0: no pain'' and ''10: worst pain'' .

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan Akkaya, Study Chair — Diskapi Yildirim Beyazıt Teaching and Research Hospital; Gevher Rabia Genç Perdecioğlu, Study Director — Diskapi Yildirim Beyazıt Teaching and Research Hospital; Hüseyin Alp Alptekin, Principal Investigator — Diskapi Yildirim Beyazıt Teaching and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazıt Teaching and Research Hospital, Ankara, Turkey (Türkiye)